CLINICAL TRIAL: NCT03184753
Title: Innovative Treatment of Ovarian Cancer Based on Immunogene-modified T Cells (IgT)
Brief Title: Genetically Modified T Cells Against Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, Principal Investigator, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17002
Record Dates: First submitted 2017-06-04; First posted 2017-06-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
Keywords: Autologous; IgT; Ovarian Cancer; CART
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): OC-IgT cells to treat ovarian cancer.
  Interventions: Biological: OC-IgT cells

INTERVENTIONS:
Biological: OC-IgT cells — Autologous human OC-IgT cells.

SUMMARY:
The primary objectives are to evaluate the safety and efficacy of infusion of autologous ovarian cancer immunogene-modified T cells (OC-IgT cells).

DETAILED DESCRIPTION:
Ovarian cancer (OC) is a cancer that forms in or on an ovary. The majority of OC arises from the epithelium (outer lining) of the ovary. In 2015 OC was found in 1.2 million women and resulted in 161,100 deaths worldwide. Among women it is the seventh-most common cancer and the eighth-most common cause of death from cancer. Treatment for OC consists of surgery, chemotherapy, radiotherapy and sometimes, novel immunotherapies. The best treatment options depend on many factors, including the type of OC, its stage and grade, as well as the general health of the patient.

Adoptive immunotherapy with cytotoxic T lymphocytes reactive with specific antigens has proven to be effective. Novel chimeric antigen receptor gene modified T cell (CART) based immunotherapy has demonstrated great successes in B cell malignancies. Here, the study aim is to evaluate the safety and efficacy of genetically engineered OC-specific and immune modulatory T cells in patients. The primary study objectives are to evaluate the safety of the investigational product, autologous OC-IgT cells, to subjects by IV and intratumoral injection. The secondary study objectives are (1) to evaluate the success rate of generating autologous OC-IgT cells in vitro, and (2) to determine the anti-OC efficacy of the OC-IgT cells.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent obtained prior to any study-specific procedures.
2. Female patients ≥ 20 years.
3. Eastern Cooperative Oncology Group (ECOG) PS of 0, 1 or 2.
4. Life expectancy ≥ 3 months.
5. Able to comply with the protocol.
6. Histologically confirmed and documented high risk International Federation of Gynecology and Obstetrics (FIGO): Stage III-IV.

   * Complete remission after salvage treatment for first recurrence.
7. Not pregnant, and on appropriate birth control if of childbearing potential.
8. Adequate bone marrow reserve with ·absolute neutrophil count (ANC) ≥ 1000/mm3.

   ·Platelets ≥100,000/mm3.
9. Adequate renal and hepatic function with ·Serum creatinine ≤ 2 x upper limit of normal (ULN). ·Serum bilirubin ≤ 2 x ULN.

   * aspartate aminotransferase (AST)/ALT ≤ 2 x ULN.
   * Alkaline phosphatase ≤ 5 x ULN.
   * Serum bilirubin. 2.0 is acceptable in the setting of known Gilbert's syndrome.

Exclusion Criteria:

1.Patients with:

* Non-epithelial ovarian cancer.
* Ovarian tumors with low malignant potential (i.e. borderline tumors).
* Synchronous primary endometrial carcinoma and ovarian cancer. 2.Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure (prior, current or planned treatment).

Previous experience of gene-engineered T cell therapy 4.Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug or previous participation in this study.

5.Minor surgical procedures within 2 days prior to Day 0 (including central venous access device placement for chemotherapy administration, tumor biopsies, needle aspirations).

6.Pregnant or lactating females. 7.Inadequate bone marrow function:

·Absolute neutrophil count < 1.0 x 109/L.

* Platelet count < 100 x 109/L.
* Hb < 9 g/dL. 8. Inadequate liver and renal function:
* Serum (total) bilirubin > 1.5 x ULN.
* AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases).
* Alkaline phosphatase > 2.5 x ULN (or > 5 x ULN in case of liver metastases or > 10 x ULN in case of bone metastases).
* Serum creatinine >2.0 mg/dl (> 177 μmol/L).
* Urine dipstick for protein uria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.

  9. Serious active infection requiring i.v. antibiotics at during screening. 10. Subject infected with HIV (HIV antibody positive), Treponema pallidum antibody positive or TB culture positive.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of adverse effects after OC-IgT cells injection | up to one month
  To assess the safety of autologous OC-IgT cells in vivo. The percentage of patients who have adverse effects will be evaluated by using the NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Rate of successful OC-IgT generation | up to one month
  The percentage of successful OC-IgT generation, which are derived from subjects and pass the safety test after standard culture procedures, viable for at least one prepatation, will be evaluated.
Ability of OC-IgT cells to induce anti-ovarian cancer reaction | after 1 month from OC-IgT cells infusion until 12 months after infusion
  measurement of CA125 concentration in blood sample
Ability of OC-IgT cells for anti-ovarian cancer reaction | after 1 month from OC-IgT cell infusion until 24 months after infusion
  Objective response (complete response (CR) + partial response (PR)) was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No